CLINICAL TRIAL: NCT07217171
Title: A Phase 1 Dose-Escalation and Expansion Study Evaluating the Safety, Efficacy, and Pharmacokinetics of EVOLVE104 in Subjects With Advanced Urothelial and Squamous Cell Carcinomas
Brief Title: A Study Evaluating the Safety, Efficacy, and Pharmacokinetics (PK) of EVOLVE104 in Participants With Advanced Urothelial and Squamous Cell Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EvolveImmune United, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EIU-104101
Record Dates: First submitted 2025-10-10; First posted 2025-10-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer; Squamous Cell Carcinoma of the Lung; Esophageal Squamous Cell Carcinoma; Tongue Squamous Cell Carcinoma; Cutaneous Squamous Cell Cancer; Penile Squamous Cell Carcinoma; Anal Squamous Cell Carcinoma; Vulvar Squamous Cell Carcinoma; Cervical Squamous Cell Carcinoma; Vaginal Squamous Cell Carcinoma; Urethral Squamous Cell Carcinoma
Keywords: bladder; lung; esophagus; tongue; penile; anal; vulvar; cervical; vaginal
MeSH Terms: conditions — Urinary Bladder Neoplasms; Esophageal Squamous Cell Carcinoma; Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1a of the study includes up to 10 participant groups given escalating dose levels of EVOLVE104 until the maximum tolerated dose(s) are reached. A Safety Review Committee will convene to review safety data from each cohort prior to dosing the next highest dose level.
  Phase 1b of the study will enroll two expansion cohorts, participants in each cohort will receive one of the selected doses from Phase 1a that may be opened at the Sponsors discretion depending on the outcome of Phase 1a. One or more doses or dose regimens of EVOLVE104 may be recommended.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Phase 1a Cohort 1; dose level 1 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 2; dose level 2 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 3; dose level 3 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 4; dose level 4 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 5; dose level 5 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 6; dose level 6 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 7; dose level 7 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 8; dose level 8 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 9; dose level 9 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1a Cohort 10; dose level 10 (Experimental): Active Study Drug
  Interventions: Drug: EVOLVE104
- Phase 1b Cohort 1; dose level TBD (Experimental): Active study drug
  Interventions: Drug: EVOLVE104
- Phase 1b Cohort 2; dose level TBD (Experimental): Active study drug
  Interventions: Drug: EVOLVE104

INTERVENTIONS:
Drug: EVOLVE104 — EVOLVE104 is provided as a solution for injection via IV infusion
  Arms: Phase 1a Cohort 10; dose level 10; Phase 1a Cohort 1; dose level 1; Phase 1a Cohort 2; dose level 2; Phase 1a Cohort 3; dose level 3; Phase 1a Cohort 4; dose level 4; Phase 1a Cohort 5; dose level 5; Phase 1a Cohort 6; dose level 6; Phase 1a Cohort 7; dose level 7; Phase 1a Cohort 8; dose level 8; Phase 1a Cohort 9; dose level 9
Drug: EVOLVE104 — Dose levels for Phase 1b will be determined based on the outcome of Phase 1a
  Arms: Phase 1b Cohort 1; dose level TBD; Phase 1b Cohort 2; dose level TBD

SUMMARY:
The goal of this study is to evaluate the safety and effectiveness of EVOLVE104 in participants with advanced urothelial and squamous cell carcinomas who have previously taken standard treatment options, have declined or have been ineligible for treatment with these medications. Participants with advanced or metastatic cancer who meet all eligibility criteria may be eligible to participate in the study.

DETAILED DESCRIPTION:
This is a dose-escalation and expansion First in Human phase 1a/1b study evaluating safety, tolerability, and pharmacokinetics (PK) of EVOLVE104 in participants with advanced, relapsed or refractory solid tumors, including bladder, lung, esophageal, tongue, cutaneous and anogenital squamous cell carcinomas. This study consists of Phase 1a dose-escalation stage followed by a Phase 1b dose expansion stage featuring 2 expansion cohorts that may be opened, at the Sponsor's discretion, depending on the safety, efficacy, and other observations from Phase 1a.

This study is anticipated to enroll approximately 160 participants: up to 80 participants in Phase 1a, and up to 80 participants in Phase 1b.

Participants will be treated until they meet treatment discontinuation criteria, including disease progression, adverse events (AEs), subject decision, investigator decision, withdrawal of consent, death. The expected duration of treatment in this study is approximately 10 months based on the anticipated progression rates for the represented malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

Participants must have locally advanced or metastatic cancer with one of the following tumor types: bladder cancer, squamous cell carcinoma of the lung, esophagus, skin, or an anogenital squamous cell carcinoma.

1. Participant must have documented disease progression during or post treatment with standard of care, dependent upon tumor type.
2. The cancer must be measurable by CT scan or MRI.
3. Eastern Cooperative Oncology Group (ECOG) performance status score ≤1.
4. Anticipated life expectancy of at least 3 months.
5. Adequate organ function, as indicated by standard blood tests.
6. Able to provide a fresh or archival tumor biopsy.
7. Male and female participants must agree to use contraception during the study and for 120 days after the last dose of study drug, except for women who are post-menopausal or surgically sterile.

Key Exclusion Criteria:

1. The participant is a candidate for treatment with a targeted agent known to provide a benefit.
2. Persistent significant toxicities from prior anticancer therapy.
3. Brain metastases unless previously treated and stable.
4. Prior severe or life-threatening immunologic reactions to previous therapies.
5. Significant medical conditions, including but not limited to:

   * History of clinically significant cardiac disease
   * Severe esophageal disease such as esophageal rupture or severe erosive esophagitis.
   * Active inflammatory corneal or conjunctival inflammation, erosion, or ulcerations.
   * History of cirrhosis or significant portal hypertension.
   * Uncontrolled or significant infection.
   * History of certain other cancers in the past 3 years.
   * History of arterial thrombosis, stroke and transient ischemic attack within 6 months.
   * Active or uncontrolled HIV, HBV or HCV infection.
   * Autoimmune or other condition requiring chronic systemic immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2029-01-29 (Estimated); Study Completion 2031-01-29 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Baseline, through study completion, an average of 10 months.
  TEAEs will be assessed during routine study visits and compared to Baseline to continuously evaluate safety and tolerability
Number of patients with Dose Limiting Toxicities (DLTs) | Baseline, through study completion, an average of 10 months.
  Protocol-defined potential DLTs will be assessed by the Safety Review Committee at routine intervals.
To determine the maximum tolerated dose (MTD) and/or recommended dose(s) for expansion (RDEs) for EVOLVE104 | Baseline, through study completion, an average of 10 months.
  Safety evaluations will occur consistently for each subject and across patients to assess MTD or RDE. Evaluations include analysis of TEAEs as well as ongoing assessments of laboratories, ECGs and physical examinations.
To determine the recommended phase 2 dose (RP2D) of EVOLVE104 | Safety evaluations will be done as described above. PK and PD to be done each cycle (28 days) at pre-dose and post dose starting Day 1 at various time points, dependent upon treatment regimen assigned, through study completion, an average of 10 months.
  Selection of the RP2D will be based on the aggregate safety, efficacy, PK, and PD observations for the entire study

SECONDARY OUTCOMES:
Assess the efficacy of EVOLVE104 | Baseline, through study completion, an average of 10 months.
  Efficacy will be evaluated through analysis of the overall response rate (ORR), including rates of complete response (CR), partial response (PR); and duration of response (DOR), and disease control rate (DCR) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
Evaluate the Cmax of EVOLVE104 | PK and PD to be done each cycle (28 days) at pre-dose and post dose starting Day 1 at various time points, dependent upon treatment regimen assigned, through study completion, an average of 10 months.
  The maximum observed plasma concentration will be evaluated.
Evaluate the Tmax of EVOLVE104 | PK and PD to be done each cycle (28 days) at pre-dose and post dose starting Day 1 at various time points, dependent upon treatment regimen assigned, through study completion, an average of 10 months.
  The duration of time taken to reach Cmax will be evaluated.
Evaluate the Area Under the Curve (AUC) for EVOLVE104 | PK and PD to be done each cycle (28 days) at pre-dose and post dose starting Day 1 at various time points, dependent upon treatment regimen assigned, through study completion, an average of 10 months.
  AUC time curve from 0 to 24 hrs post dose and percent difference between intervals will be evaluated.
Evaluate the incidence of anti-drug antibodies (ADA) to EVOLVE104 | Collected pre-dose cycle 1 and then every other cycle starting with cycle 4
  The presence of ADAs and their clinical impact will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: EvolveImmune Study Team, Study Director — EvolveImmune United, Inc
Locations (5):
- United States (5):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - The Winship Cancer Institute Emory University, Atlanta, Georgia
  - START Midwest, Grand Rapids, Michigan
  - SCRI, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia